CLINICAL TRIAL: NCT04866043
Title: Drug Utilization Study With VYVANSE® in Australia for Binge Eating Disorder
Brief Title: Drug Use Study With VYVANSE® in Australia for Binge Eating Disorder
Status: Completed | Type: Observational
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: SHP489-827; EUPAS40690 (Registry Identifier: EU PAS Register)
Record Dates: First submitted 2021-04-28; First posted 2021-04-29 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Binge-eating Disorder
MeSH Terms: conditions — Binge-Eating Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NostraData Database: All prescriptions for lisdexamfetamine dimesylate available in the NostraData database at any time in the last 12 months will be collected in Australia.
- Physician Survey: Physician will provide de-identified data of participants who have been prescribed lisdexamfetamine dimesylate at least once during the study period for indications other than attention deficit hyperactivity disorder (ADHD) in Australia.

SUMMARY:
This study will check how and to whom Vyvanse is prescribed in Australia by retrospectively analyzing a prescription database with additional information provided by a physician survey.

DETAILED DESCRIPTION:
This is a drug utilization study (DUS) using cross-sectional database analysis of participants who are prescribed lisdexamfetamine dimesylate for treatment of BED. The study will combine data from two sources of patient-level drug utilization data for lisdexamfetamine dimesylate:

* NostraData database: Longitudinal participant level prescription dispensing database
* Physician survey: De-identified participant data provided by representative psychiatrists and other physicians expected to treat participants with BED in Australia.

In the NostraData database, actual drug dispensing data are collected, which allows for the generation of information on actual drug usage. However, these data do not contain certain participant variables, such as age and indication, needed to monitor potential off-label use. Therefore, these data must be supplemented with another data source. The physician survey will provide the data not included in the NostraData database.

The DUS will enroll approximately 150 participants.

This DUS will be conducted in Australia. The overall time for data collection in the study will be approximately 36 months after the launch date of lisdexamfetamine dimesylate.

ELIGIBILITY:
Inclusion Criteria:

Main prescription data analysis:

- At least one prescription for lisdexamfetamine dimesylate recorded in the NostraData database in Australia.

For all sensitivity analyses (sensitivity analysis I, II and III):

- At least one prescription for lisdexamfetamine dimesylate recorded in the NostraData database in Australia during the defined observation period of the study.

Physician survey:

- The physician prescribed lisdexamfetamine dimesylate for indications other than ADHD in the last 12 months for at least one participant.

Participant population:

- Physician entered data for the participant until at least question 3 (treatment information (Q03); main indication).

Exclusion Criteria:

For all sensitivity analyses (sensitivity analysis I, II and III):

* Evidence of use for lisdexamfetamine dimesylate for treatment of ADHD, as shown by prescription records for ADHD medication other than lisdexamfetamine dimesylate at any time.
* Record of at least one lisdexamfetamine dimesylate prescription prior to launch of lisdexamfetamine dimesylate for BED (02/17/2018).

Additional exclusion criteria for the specific sensitivity analyses:

For sensitivity analysis I:

- Prescriptions for lisdexamfetamine dimesylate issued by pediatricians or child psychiatrists.

For sensitivity analysis II:

- Prescriptions for lisdexamfetamine dimesylate issued by all prescribers other than psychiatrists (example, pediatricians, general practitioner [GPs]).

For sensitivity analysis III:

* Prescriptions for lisdexamfetamine dimesylate issued by pediatricians or child psychiatrists.
* For participants with age available, participants with evidence for age at first prescription below 18 years.

Physician survey and participant population:

- Physician entered ADHD as main indication for prescription of lisdexamfetamine dimesylate (treatment information [Q03]) for the participant.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants who have been prescribed lisdexamfetamine dimesylate at least once during the reporting period without evidence of use of lisdexamfetamine dimesylate for ADHD treatment.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Number of Participants Based on Indication of Use of Lisdexamfetamine Dimesylate | Up to 36 months
  Number of participants based on indication of use of Lisdexamfetamine Dimesylate will be assessed.

SECONDARY OUTCOMES:
Number of Participants Based on Patterns of Drug Use | Up to 36 months
  Number of participants based on patterns of drug use will be assessed.
Number of Participants Based on Average Daily Dose | Up to 36 months
  Number of participants based on average daily dose will be assessed.
Number of Participants Based on Maximum Daily Dose | Up to 36 months
  Number of participants based on maximum daily dose will be assessed.
Number of Participants Based on Co-prescription | Up to 36 months
  Number of participants based on co-prescription of lisdexamfetamine dimesylate with monoamine oxidase inhibitors (MAOIs), selective serotonin reuptake inhibitors (SSRIs), serotonin-norepinephrine reuptake inhibitors (SNRIs), guanfacine hydrochloride and other central nervous system (CNS) stimulants will be assessed.
Number of Participants Based on Co-diagnosis | Up to 36 months
  Number of participants based on co-diagnosis (BED and other indications except ADHD) will be assessed.
Number of Prescriptions of Lisdexamfetamine Dimesylate | Up to 36 months
  Number of Prescriptions of lisdexamfetamine dimesylate will be evaluated.
Treatment Duration | Up to 36 months
  Treatment duration will be defined as the length of time a participant remains on treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (1):
- Site, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/60901ad9f89629001e47b504